CLINICAL TRIAL: NCT04782427
Title: COVID-19 Infections and Mortality in Montreal Long-term Care Facilities During the First Wave: a Retrospective Cohort Study
Brief Title: COVID-19 Infections and Mortality in Long-term Care Facilities During the First Wave
Status: Completed | Type: Observational
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Collaborators: Université de Montréal (Other)
Responsible Party: Principal Investigator, Sophie Zhang, Head physician of long-term care facilities and researcher, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Other Study IDs: CentreSuddeMontréal
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Covid19; Death; Infection Viral; Infections, Respiratory; Infection, Coronavirus; Elderly Infection; Old Age; Dementia; Epidemic Disease
MeSH Terms: conditions — COVID-19; Death; Virus Diseases; Respiratory Tract Infections; Coronavirus Infections; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: COVID-19 infection — Case of nosocomial infection within the long-term care facility

SUMMARY:
The medical charts of all COVID-19 cases (n=1200) from 17 long-term care facilities in Montreal, Canada will be reviewed, to compare patients who survived to patients who did not survive. Through multilevel logistic regression, the risk of death will be estimated for institutional predictors of mortality, while controlling for individual risk factors.

Individual covariates include clinical features (age, sex, Charlston comorbidity index, SMAF autonomy score, severity criteria) and medical treatments (IV fluids, anticoagulation, oxygen, regular opiates, corticosteroids). Aggregate covariates include epidemiological data (attack rates, timing of outbreak) and institutional characteristics (number of beds, air exchange per hour, presence of a dedicated COVID-19 unit at the time of outbreak, staff compliance to infection control measures, staff infection rates, understaffing, proportion of semi-private rooms, proportion of wandering wards and other special units).

DETAILED DESCRIPTION:
A lot has been written about individual risk factors for COVID-19 death, mostly in the hospitalized population. However, even though most deaths around the world have occurred among the frail and elderly, little is known about the risk factors specific to the long-term care population.

In this retrospective cohort study, the investigators will review the medical charts of all COVID-19 cases (n=1200) from 17 long-term care facilities in Montreal, Canada, to compare patients who survived to patients who did not survive. Through multilevel logistic regression, the risk of death will be estimated for institutional predictors of mortality, while controlling for individual risk factors. The objective is to influence local and national policies in long-term care facilities, in the hopes of avoiding the tragic spring 2020 outcomes during subsequent waves of COVID-19 or future pandemics.

Covariates in the models will be drawn from a review of the medical literature and known risk factors for COVID-19 death. Individual-level covariates include clinical features (age, sex, Charlston comorbidity index, SMAF autonomy score, severity criteria) as well as medical treatments (IV fluids, anticoagulation, oxygen, regular opiates, corticosteroids). Aggregate-level covariates include epidemiological data (attack rates, timing of outbreak) and institutional characteristics (number of beds, air exchange per hour, presence of a dedicated COVID-19 unit at the time of outbreak, staff compliance to infection control measures, staff infection rates, understaffing, proportion of semi-private rooms, proportion of wandering wards and other special units).

ELIGIBILITY:
Inclusion Criteria:

* Resident of a long-term care facility within the CIUSSS Centre-Sud-de-l'Île-de-Montréal
* Nosocomial COVID-19 infection diagnosis between March 23rd and July 11th 2020

Exclusion Criteria:

* Admission to the long-term care facility after July 11th 2020
* COVID-19 infection which was not acquired within the long-term care facility

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Most of the residents living in the long-term care facilities are elderly and frail, with a high prevalence of major neurocognitive disorders and low life expectancy. However, some patients are more robust (e.g. residents of wandering wards) or younger (e.g. residents with heavy neurological or mental health diagnoses).
Sampling Method: Probability Sample
Enrollment: 1197 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-05-13 (Actual)

PRIMARY OUTCOMES:
Death | 28 days
  COVID-19 as a primary or secondary cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Zhang, M.D., Principal Investigator — Université de Montréal
Locations (1):
- CIUSSS Centre-Sud-de-l'Île-de-Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All deidentified information will be shared, except if there are patient confidentiality issues.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the time of publication, for 5 years.
Access Criteria: Written request submitted to the principal investigator.